CLINICAL TRIAL: NCT04816032
Title: "Effectiveness of the Expressive Writing on the Somatization and Psychological Health of the Migrants: a Longitudinal Study"
Brief Title: "Expressive Writing Psychological Health Migrants (EWPHM)
Acronym: EWPHM
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Roma La Sapienza (Other)
Responsible Party: Principal Investigator, Carlo Lai, Associate Professor, University of Roma La Sapienza
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: URomLS_3
Record Dates: First submitted 2021-03-18; First posted 2021-03-25 (Actual); Last update posted 2021-03-30 (Actual); Status verified 2021-03

CONDITIONS: Psychological Health
Keywords: expressive writing treatment psychological health migrants
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Pennebaker's expressive writing (Experimental): Three consecutive days for 20 minutes daily of expressive writing. The topic of the traumatic traveling experience, focalizing the attention on the deeper emotions, thoughts, and feelings.
  Interventions: Other: Pennebaker's expressive writing intervention
- Writing about different aspects of their knowledge (Active Comparator): Three consecutive days for 20 minutes daily of neutral writing. Different topics of own knowledge Description of the city, their room, their place where they live, or easy procedure like, how to make a coffee (or something else), their population, trying to remain free from deep emotions, thoughts, or feelings.
  Interventions: Other: Neutral writing
- Control (No Intervention): No intervention

INTERVENTIONS:
Other: Pennebaker's expressive writing intervention — It focuses on the emotional aspect of the written event
  Arms: Pennebaker's expressive writing
Other: Neutral writing — Description of neutral topics with less emotional involvement
  Arms: Writing about different aspects of their knowledge

SUMMARY:
Migration is a global phenomenon that produces several psychological impacts on the migrant causing psychological changes and difficulties such as the development of psychological diseases, the decrease of the life expectancy, insecurity, isolation, and poorness. These diseases create a situation of emergency that has prompted the need to intervene with specific psychological treatments. This study proposed to verify the effectiveness of expressive writing on the elaborative processes of the migratory journey's trauma. Participants were twenty-eight migrants of a reception center. A blinded randomized controlled trial was performed to divide them into three groups: an experimental sample that performed the expressive writing treatment, a neutral sample that performed the neutral description writing, and a control sample. The samples were assessed in three times through self-report measures. The administration of expressive writing is expected to improve the psychological health condition of migrants

DETAILED DESCRIPTION:
Emigration is a global phenomenon with a significant impact in both, host countries and especially on people who decide to migrate. Italy seems to be a chosen destination for migrants, mainly due to its geographical position, as one of the European Union's border countries. Italy is mentioned as the fifth European country in Europe about the number of migrants. Currently, there are 5 million immigrants in Italy. Recent migratory flows in Italy have changed the cultural background of the main communities residing in the country. However, several studies have pointed out that the migration phenomenon is not a comfortable linear process, on the contrary, there are difficulties related to migratory traveling and the way it is carried out. Among others, the traveling experience could leave relevant marks on a psychological level. Recent studies underlie the effect of migration on the development of psychological diseases, on the loss of hope for the future that it affected the life expectancy causing insecurity, isolation, and poorness, and producing modification on the possible existing symptomatology. Moreover, the discrimination and disorientation that migrants experience while traveling and in host countries seem to have a relationship with anxiety symptoms.

Therefore, many investigations applied psychological intervention to treat the described symptomatology. The literature highlights the importance of the treatments such as cognitive-behavioral therapy, narrative exposure therapy, dynamic therapy, combined psychological treatments, and combined psychological with pharmacological treatments. Of the mentioned treatments, the narrative exposure treatment seems to be the less applied intervention, a meta-analysis suggested a fairly effective application of NET on populations with trauma, however, this result must be taken with caution. The NET is a trauma-focused therapy, based on trauma expositions in an autobiographical context. This treatment provides both verbal and non-verbal application, as the expressive writing-EW. Additionally, Pennebaker considered that expressive writing referring to the own traumatic events with emotional descriptions could be of help in the resolution of the own life narrations and the insert of own memories in life history. The expressive writing technique applies to the own serious traumatic events, from 3 to 5 consecutive days, for 15 minutes daily. This technique is more structured compare to NET which can be both written and oral and doesn't necessarily provide a brief exposition. The expressive writing is applied in a more extended context of trauma, violence, war, natural catastrophe, cancer, and torture. Currently in literature, there not seem to be any authoritative studies that have applied the expressive writing technique to the trauma of the migratory journey. The present investigation allows extending the acknowledgment of this treatment applied to a population of adult migrants submitted to forced migration.

The aim of this study was to provide evidence of the effectiveness of expressive writing on mental and physical health in migrants considering the mediation role of the hope for the future. The hypothesis was that migrants who performed an expressive writing treatment will show a decrease in symptomatology in association with a greater sense of hope for the future.

The study involved three different samples: experimental, neutral, and control group. The three samples were composed through a randomized controlled trial placing 22 participants for each sample. The random allocation of participants within the three samples was blindly performed.

The non-profit association "Medihospes" located in Rome provided the migrant participants. Each participant was invited to read and accept the study by completing and signing the informed consent form. The inclusion criteria were age >18 years and the refugees' or asylum seekers' status. The exclusion criteria were psychiatric or neurologic diagnosis and drug abuse.

The study was settled in three different times. At T0 time were administered a self-report questionnaires' battery composed of four measures: Beck Hopelessness Scale, BHS, Toronto Alexithymia Scale 20, TAS-20, Symptom Check-List Revised, SCL-90-R, Impact of Event Scale-Revised, IES-R.

After this first assessment, the participants of the experimental sample received the expressive writing Pennebaker's treatment, the participants of the neutral sample received instructions of writing on a general topic of their choice and the participants of the control sample received no treatment or instructions.

After one week to the treatment phase (T1) and after one month from T1 time (T2) the same self-report questionnaire's battery was administered to all the participants.

Treatment Pennebaker's expressive writing was applied for three consecutive days for 20 minutes daily. The participants of the experimental sample were asked to write about the traumatic traveling experience, focalizing the attention on the deeper emotions, thoughts, and feelings.

The participants of the neutral sample were asked to write about different topics of their knowledge for three consecutive days for 20 minutes daily; the topics could relate the description of the city, their room, their place where they live, or easy procedure like, how to make a coffee (or something else), or to describe their population, trying to remain free from deep emotions, thoughts or feelings.

ELIGIBILITY:
Inclusion Criteria:

* age >18 years and the refugees or asylum seekers status

Exclusion Criteria:

* psychiatric or neurologic diagnosis and drug abuse.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2017-11-02 (Actual); Primary Completion 2018-03-15 (Actual); Study Completion 2018-07-30 (Actual)

PRIMARY OUTCOMES:
psychological health of the migrants assessed with Symptom Check-List Revised. A self-report questionnaire that assess the psychological and psychopathological dimensions | 1 month
  Specifically, the somatization and in general, the global psychological functioning. The Symptom Check-List Revised Scale was a self-report questionnaire that measures psychological and psychopathological issues in clinical and non-clinical populations. It is composed from 90 items. Higher scores show the presence of psychopathological symptomology and psychological complications. The range of scores are less 45 more 75 with cut-off 55. It is composed by different dimensions.

SECONDARY OUTCOMES:
Hope for the future, assessed with Beck Hopelessness Scale, self-report questionnaire | 1 month
  The outcome was assessed with Beck Hopelessness Scale. The scale is a self-report that quantifiy the hopelessness within three specific subscales (future, motivation, and expectation). Higher score means higher greater loss of hope for the future. The range of the scores are 0-20 with cut-off 9 (moderate loss of hope)

CONTACTS AND LOCATIONS:
Overall Officials: Carlo Lai, Professor, Principal Investigator — University of Roma La Sapienza
Locations (2):
- Italy (2):
  - Carlo Lai Professor PhD, Roma, Rm
  - Department of Dynamic and Clinical Psychology, and Health Studies, Sapienza University, Rome

IPD SHARING:
Plan to Share IPD: Yes
The data was collected and stored by the Dynamics department and clinical psychology laptop, protected by a password. The data are accessible only to the Chief Researcher, the Ph.D. student, and the secondary researcher. The study protocol will be shared with other sub-investigators involved in the study, but not sensitive data. The study report will be shared and published in a scientific journal, but the privacy of each participant will be respected according to the agreements established by the ethics committee.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: 24 months
Access Criteria: The sensitive data are collected in an excel database on the department of Dynamic and Clinical psychology laptop, protected by a password. Each participant is identified by a personal numerical code, to guarantee them their privacy. All the sensitive data will be accessible only by the Chief investigator, the Ph.D. student, and the sub-investigator co-responsible for the study

REFERENCES:
- [Derived] Begotaraj E, Sambucini D, Ciacchella C, Pellicano GR, Pierro L, Wamser-Nanney R, Aceto P, De Paola C, Caroppo E, Lai C. Effectiveness of the expressive writing on the psychological distress and traumatic symptoms of the migrants: A prospective study multiarm randomized controlled trial. Psychol Trauma. 2023 Jul;15(5):738-747. doi: 10.1037/tra0001308. Epub 2022 Sep 29. PMID 36174151